CLINICAL TRIAL: NCT07298421
Title: A Phase III Randomized Double-Blind Multi-Center Treat-Through Study to Evaluate the Pharmacokinetics, Safety and Efficacy of Induction and Maintenance Therapy With Afimkibart (RO7790121) in Children Aged 2-17 Years With Moderately to Severely Active Crohn's Disease
Brief Title: A Study to Assess the Pharmacokinetics, Effectiveness and Safety of Afimkibart for Induction and Maintenance Therapy in Children With Moderately to Severely Active Crohn's Disease
Acronym: SIBERITE-PEDS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP45906; 2025-523318-96-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-19; First posted 2025-12-23 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Moderately to Severely Active Crohns Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Afimkibart Dose A (Experimental): Participants will receive Afimkibart intravenously (IV) followed by Afimkibart subcutaneous (SC) injection.
  Interventions: Drug: Afimkibart
- Afimkibart Dose B (Experimental): Participants will receive Afimkibart IV followed by Afimkibart SC.
  Interventions: Drug: Afimkibart

INTERVENTIONS:
Drug: Afimkibart — Afimkibart will be administered as IV infusion. Afimkibart will be administered as SC injection.
  Other Names: RO7790121; PF-06480605; RVT-3101

SUMMARY:
This phase III, double-blind, multi-center treat-through study will evaluate the efficacy and safety of Afimkibart (also known as RO7790121) in children with moderately to severely active Crohn's Disease (CD).

ELIGIBILITY:
Inclusion Criteria:

* Body weight >= 10 kilogram (kg)
* Active CD confirmed by endoscopy (ileocolonoscopy)
* Moderately to severely active CD, defined as a Pediatric Crohn's Disease Activity Index (PCDAI) score >= 30, and Simple Endoscopic Score Crohn's Disease (SES-CD) >=6 (or >=4 for isolated ileal disease) confirmed through centrally-read ileocolonoscopy
* Inadequate response, loss of response, and/or intolerance to at least one of the following conventional therapies (aminosalicylates, corticosteroids and/or immunosuppressants) or advanced therapies (including anti-tumor necrosis factor, anti-interleukin, anti-integrin, or Janus Kinase (JAK) inhibitors)

Exclusion Criteria:

* Monogenic disorder pertaining to infant onset Inflammatory Bowel Disease (IBD)
* History of >= 3 bowel resections: > 2 missing segments of the following five segments: terminal ileum, right colon, transverse colon, sigmoid and left colon, and rectum
* Current diagnosis of ulcerative colitis (UC), abdominal/intraabdominal/perianal fistula and/or abscess, indeterminant colitis, IBD-unclassified, microscopic colitis, ischemic colitis, infectious colitis, radiation colitis, or active diverticular disease.
* Symptomatic bowel strictures, fulminant colitis, or toxic megacolon
* Presence of abdominal or perianal abscess
* Current diagnosis or suspicion of primary sclerosing cholangitis

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2026-05-29 (Estimated); Primary Completion 2030-05-29 (Estimated); Study Completion 2031-05-29 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Clinical Remission per Pediatric Crohn's Disease Activity Index (PCDAI) | At Week 52
Percentage of Participants With Endoscopic Response | At Week 52

SECONDARY OUTCOMES:
Percentage of Participants With Clinical Remission | At Week 12 and Week 52
Percentage of Participants With Clinical Response | At Week 12 and Week 52
Percentage of Participants With CDAI Remission | At Week 12 and Week 52
Change From Baseline in Fecal Calprotectin | Baseline, Week 12 and Week 52
Change From Baseline in Mucosal Inflammation Noninvasive Index (MINI) Score | Baseline, Week 12 and Week 52
Percentage of Participants With Endoscopic Remission | At Week 52
Percentage of Participants With Corticosteroid-Free Clinical Remission | At Week 52
Percentage of Participants with Maintenance of Remission | At Week 12 and Week 52
Percentage of Participants With Histologic Improvement | At Week 52
Percentage of Participants With Ulcer-Free Endoscopy | At Week 52
Incidence and Severity of Adverse Events (AEs) | Up to Approximately 5.5 Years
Serum Concentration of Afimkibart | Up to Approximately 5.5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing